CLINICAL TRIAL: NCT05172284
Title: Registry and Monitoring of ImmuNe-mediated Inflammatory Diseases (IMIDs) REMIND Study
Brief Title: Registry and Monitoring of ImmuNe-mediated Inflammatory Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: REMIND
Record Dates: First submitted 2021-12-09; First posted 2021-12-29 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: ImmuNe-Mediated Inflammatory Diseases
MeSH Terms: interventions — Surveys and Questionnaires; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Psoriasis
  Interventions: Other: Questionnaires
- Psoriatic arthritis
  Interventions: Other: Questionnaires
- Atopic dermatitis
  Interventions: Other: Questionnaires
- Chronic urticaria
  Interventions: Other: Questionnaires
- Suppurative hydrosadenitis
  Interventions: Other: Questionnaires
- Systemic lupus erythematosus
  Interventions: Other: Questionnaires
- Acne vulgaris
  Interventions: Other: Questionnaires
- Rosacea
  Interventions: Other: Questionnaires
- Seborrheic dermatitis
  Interventions: Other: Questionnaires
- Contact dermatitis
  Interventions: Other: Questionnaires
- Chronic eczema of the hands
  Interventions: Other: Questionnaires
- Vitiligo
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — This is a collection of data from normal clinical routine: patients will be asked to record the assessments they undergo during their course of treatment, without changing clinical practice in any way. Data inherent to the following procedures will be collected: examinations, laboratory tests, imaging tests, questionnaires and rating scales.
  Other Names: blood tests; instrumental and/or imaging examinations; rating scales

SUMMARY:
Formation of a registry of IMID patients to assess the evolution of resistance to conventional and target therapies. This aim is achieved by evaluating the achievement of PASI 50 and PASI 75 scores at week 16 from the start of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of IMID.
* Patients of any age, including minors.
* Patients treated with approved medications for the condition in question and/or phototherapy.
* Patients who agree to sign informed consent.

Exclusion Criteria:

* Patients without a diagnosis of IMID.
* Patients who do not consent to sign informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In this study (registry) will be included all IMID patients afferent to the UO of Dermatology of IRCCS Istituto Ortopedico Galeazzi for an estimated total of 5 years of recruitment.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Registry of ImmuNe-mediated inflammatory Diseases (IMIDs) | 15 years
  Formation of a registry of IMID patients to assess the evolution of resistance to conventional and target therapies.

SECONDARY OUTCOMES:
PASI 50 | 15 years
  Assess attainment of PASI 50 score from the start of treatment to all follow-ups
PASI 75 | 15 years
  Assess attainment of PASI 75 score from the start of treatment to all follow-ups

OTHER OUTCOMES:
Special populations | 15 years
  Quantification and monitoring of IMID patients belonging to "special populations". Special populations include: homeless, transgender, amputees, para and quadriplegics.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Damiani, Dr., Principal Investigator — IRCSS Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No